CLINICAL TRIAL: NCT06700941
Title: Impact of HPV Vaccination Against Cervical Lesions and Genital Warts in Colombia. an Ecological Assessment
Status: Completed | Type: Observational
Sponsor: Universidad Nacional de Colombia (Other)
Collaborators: MSD Pharmaceuticals LLC (Industry)
Responsible Party: Principal Investigator, Fernando Pio De La Hoz Restrepo, Professor, Universidad Nacional de Colombia
Other Study IDs: B.FM.1.002- CE-155-24
Record Dates: First submitted 2024-10-28; First posted 2024-11-22 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-10

CONDITIONS: Cervical Intraepithelial Neoplasia (CIN); Genital Warts; Papillomavirus Infections; Cervical Cancers
Keywords: HPV Vaccination; Cervical Intraepithelial Neoplasia; Genital warts; Preneoplastic Lesions; Human Papillomavirus
MeSH Terms: conditions — Uterine Cervical Dysplasia; Condylomata Acuminata; Papillomavirus Infections; Uterine Cervical Neoplasms | interventions — Papillomavirus Vaccines

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Vaccinated female cohort (1996-2003): This group consists of female participants born between 1996 and 2003 who were eligible for HPV vaccination starting in 2012 as part of the national immunization program in Colombia. These individuals received the vaccine and are being monitored for trends in healthcare service usage related to genital warts and preneoplastic cervical lesions.
  Interventions: Biological: HPV vaccine
- Unvaccinated Female Cohort (Before 1996): This group includes female participants born before 1996 who were not part of the HPV vaccination program. They serve as a comparison group to assess trends in healthcare service usage for genital warts and preneoplastic cervical lesions before the implementation of the HPV vaccination program.

INTERVENTIONS:
Biological: HPV vaccine — The intervention of interest in this observational study is the HPV vaccine, which was introduced as part of Colombia's national immunization program in 2012. The vaccine is administered to girls between the ages of 9 and 17 to prevent cervical cancer, preneoplastic cervical lesions, and genital warts caused by HPV infection. The vaccine schedule typically includes two doses given over six months.
  This study does not involve administering the vaccine as part of the research. Instead, it retrospectively analyzes the healthcare records of individuals who received the vaccine as part of routine care and compares outcomes with those who were not vaccinated.
  Groups: Vaccinated female cohort (1996-2003)

SUMMARY:
The goal of this observational study is to assess the impact of HPV vaccination on cervical lesions and genital warts in Colombian birth cohorts. The study examines the trends in healthcare services usage related to these conditions, particularly among vaccinated and unvaccinated populations.

The main questions it aims to answer are:

Have health services usage rates for preneoplastic cervical lesions and genital warts decreased among cohorts of girls eligible for HPV vaccination after the vaccine's introduction? Have there been reductions in health services usage for genital warts among male cohorts of the same birth years as vaccinated girls? Researchers will compare health services usage trends between vaccinated and unvaccinated populations, as well as geographical areas with differing levels of HPV vaccination coverage, to evaluate the impact of the HPV vaccination program.

Participants will not be directly involved, as this is a retrospective analysis of existing healthcare records from various national databases, assessing the frequency of healthcare services related to preneoplastic lesions and genital warts, as well as vaccination coverage at national, departmental, and municipal levels.

DETAILED DESCRIPTION:
This study is an observational ecological assessment aimed at evaluating the impact of the HPV vaccination program on the incidence of cervical preneoplastic lesions and genital warts in Colombia. The analysis compares trends in health services usage across different birth cohorts of girls and boys, exposed and unexposed to the HPV vaccine, using secondary data sources such as the National Health Service Records (UPC) and individual healthcare provision records (RIPS).

The study will employ a retrospective time-series analysis, assessing the frequency of healthcare encounters related to the targeted conditions (genital warts and preneoplastic lesions) by birth cohort and vaccination status. The primary objective is to determine whether there has been a significant reduction in healthcare service use for these conditions following the introduction of the HPV vaccine in 2012.

Secondary objectives include evaluating geographical variations in HPV vaccine coverage at the departmental and municipal levels and their association with the trends in healthcare service usage. This will help ascertain if higher vaccine coverage corresponds to lower rates of genital warts and preneoplastic cervical lesions.

The analysis will rely on both temporal (longitudinal) and geographical (cross-sectional) comparisons. Temporal trends will examine changes before and after the vaccine's introduction, while geographical analysis will compare regions based on varying vaccination coverage levels. Exposure will be categorized according to birth cohort (girls born between 1996 and 2003) and vaccination rates in different geographical areas.

The data analysis will include calculating the average annual rates of healthcare service utilization for both genital warts and preneoplastic lesions, stratified by sex, age group, and region. Statistical methods such as incidence rate ratios (IRRs) and 95% confidence intervals will quantify the association between HPV vaccination and healthcare service usage. The study will also assess potential biases, including information bias due to variability in diagnosis and reporting practices across different health service providers.

By utilizing existing records and implementing robust statistical approaches, the study aims to contribute valuable insights into the effectiveness of HPV vaccination in a middle-income country, where cervical cancer prevention strategies are not as comprehensive as in high-income countries.

The study is anticipated to run for one year, with results presented to both scientific audiences and health policy decision-makers to support the optimization of HPV vaccination strategies in Colombia.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be born between 1996 and 2003 (for vaccinated cohorts).
* Participants born before 1996 (for unvaccinated cohorts) may be included as control groups.
* Participants must have healthcare service records available for analysis related to genital warts or preneoplastic cervical lesions.
* Participants must have received or not received the HPV vaccine, according to the national immunization program records.
* Data must be available for individuals from regions with documented HPV vaccination coverage rates (departments or municipalities).

Exclusion Criteria:

* Participants without available healthcare service records for genital warts or preneoplastic cervical lesions.
* Participants with incomplete or inaccurate vaccination records.
* Participants not born within the specified birth cohort ranges (i.e., after 2003 or before 1996).
* Individuals from regions without accessible data on HPV vaccination coverage.

Ages: 9 Years to 23 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of individuals from various regions of Colombia, specifically focusing on birth cohorts from 1996 to 2003 for vaccinated groups and cohorts born before 1996 for unvaccinated groups. Participants are drawn from nationwide healthcare service utilization records (UPC and RIPS databases) and HPV vaccination records maintained by the national immunization program. The population includes both males and females, with data sourced from both urban and rural areas, covering all geographical regions with documented HPV vaccination coverage.
Sampling Method: Non-Probability Sample
Enrollment: 8000000 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Healthcare Service Usage for Genital Warts | January 1, 2012, to December 31, 2019, assessed annually.
  The primary outcome measure is the annual rate of healthcare service usage related to genital warts among vaccinated versus unvaccinated individuals. This will be assessed using healthcare service utilization records and rates will be compared across vaccinated and unvaccinated birth cohorts.
Change in Healthcare Service Usage for Preneoplastic Cervical Lesions | January 1, 2012, to December 31, 2019, assessed annually.
  The primary outcome measure is the annual rate of healthcare service usage related to preneoplastic cervical lesions among vaccinated and unvaccinated female cohorts. This measure will utilize healthcare records to assess changes in service usage over time between cohorts.

SECONDARY OUTCOMES:
Correlation between HPV Vaccination Coverage and Service Usage | January 1, 2012, to December 31, 2019, assessed annually, stratified by geographical regions.
  The secondary outcome measure assesses whether regions with higher HPV vaccination coverage have lower rates of healthcare service usage for genital warts and preneoplastic cervical lesions.
Gender-Specific Trends in Service Usage | January 1, 2012, to December 31, 2019, assessed annually.
  Assess whether there is a reduction in healthcare service usage for genital warts among males in vaccinated vs. unvaccinated birth cohorts.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Nacional de Colombia, Bogotá, Bogota D.C., Colombia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Read TR, Hocking JS, Chen MY, Donovan B, Bradshaw CS, Fairley CK. The near disappearance of genital warts in young women 4 years after commencing a national human papillomavirus (HPV) vaccination programme. Sex Transm Infect. 2011 Dec;87(7):544-7. doi: 10.1136/sextrans-2011-050234. Epub 2011 Oct 4. PMID 21970896
- [Background] Goss PE, Lee BL, Badovinac-Crnjevic T, Strasser-Weippl K, Chavarri-Guerra Y, St Louis J, Villarreal-Garza C, Unger-Saldana K, Ferreyra M, Debiasi M, Liedke PE, Touya D, Werutsky G, Higgins M, Fan L, Vasconcelos C, Cazap E, Vallejos C, Mohar A, Knaul F, Arreola H, Batura R, Luciani S, Sullivan R, Finkelstein D, Simon S, Barrios C, Kightlinger R, Gelrud A, Bychkovsky V, Lopes G, Stefani S, Blaya M, Souza FH, Santos FS, Kaemmerer A, de Azambuja E, Zorilla AF, Murillo R, Jeronimo J, Tsu V, Carvalho A, Gil CF, Sternberg C, Duenas-Gonzalez A, Sgroi D, Cuello M, Fresco R, Reis RM, Masera G, Gabus R, Ribeiro R, Knust R, Ismael G, Rosenblatt E, Roth B, Villa L, Solares AL, Leon MX, Torres-Vigil I, Covarrubias-Gomez A, Hernandez A, Bertolino M, Schwartsmann G, Santillana S, Esteva F, Fein L, Mano M, Gomez H, Hurlbert M, Durstine A, Azenha G. Planning cancer control in Latin America and the Caribbean. Lancet Oncol. 2013 Apr;14(5):391-436. doi: 10.1016/S1470-2045(13)70048-2. PMID 23628188
- [Background] Lehtinen M, Lagheden C, Luostarinen T, Eriksson T, Apter D, Harjula K, Kuortti M, Natunen K, Palmroth J, Petaja T, Pukkala E, Siitari-Mattila M, Struyf F, Nieminen P, Paavonen J, Dubin G, Dillner J. Ten-year follow-up of human papillomavirus vaccine efficacy against the most stringent cervical neoplasia end-point-registry-based follow-up of three cohorts from randomized trials. BMJ Open. 2017 Aug 18;7(8):e015867. doi: 10.1136/bmjopen-2017-015867. PMID 28821519
- [Background] Simas C, Munoz N, Arregoces L, Larson HJ. HPV vaccine confidence and cases of mass psychogenic illness following immunization in Carmen de Bolivar, Colombia. Hum Vaccin Immunother. 2019;15(1):163-166. doi: 10.1080/21645515.2018.1511667. Epub 2018 Sep 7. PMID 30118381
- [Background] la Hoz Restrepo F, Guzman NA, la Hoz Gomez A, Ruiz C. Policies and processes for human papillomavirus vaccination in Latin America and the Caribbean. Rev Panam Salud Publica. 2017 Dec 20;41:e124. doi: 10.26633/RPSP.2017.124. eCollection 2017. PMID 31391830
- See also: World Health Organization (WHO) - Human Papillomavirus (HPV) and Cervical Cancer — https://www.who.int/news-room/fact-sheets/detail/human-papillomavirus-(hpv)-and-cervical-cancer
- See also: Colombian Ministry of Health - National Immunization Program — https://www.minsalud.gov.co
- See also: National Library of Medicine (NLM) PubMed - Research Articles on HPV — https://pubmed.ncbi.nlm.nih.gov